CLINICAL TRIAL: NCT02040181
Title: Establishment of a Creatinine Clearance Estimation Equation and Daily Creatinine Excretion Reference Table for Taiwanese
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201311047RINC
Record Dates: First submitted 2013-12-22; First posted 2014-01-20 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Estimated Creatinine Clearance
Keywords: renal function, creatinine clearance

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It's important to dose according to renal function in who has impaired kidney function. There are two common methods estimating renal function: one is creatinine clearance estimated by Cockcroft-Gault (CG) equation; another is glomerular filtration rate estimated by Modification of Diet in Renal Disease (MDRD) equation.

The previous study (not published) showed that CG underestimated 24 hour measured urine creatinine clearance by our team. The difference may be due to ethnicity. Thus we want to establish a estimated creatinine clearance equation fitting in Taiwanese.

Besides, there are lots of studies discussing difference between CG and MDRD. We have found that MDRD overestimated CG in patients who were older or thin. Therefore, we want to analysis which characteristics of patients the difference are largest or smallest.

ELIGIBILITY:
Inclusion Criteria:

* age above or equal to 20 year-old adults
* had 24 hour urine creatinine collection

Exclusion Criteria:

* lack of at least one :sex, diagnosis, age,weight, height
* serum creatinine beyond linear test range
* with extreme weight or height
* with acute kidney injury or specific diagnosis
* with extremities of daily urine creatinine excretion

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients or inpatients of National Taiwan University Hospital who had 24 hour urine creatinine collections during 2010/1/1 to 2012/12/31.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Coefficient of determination of estimated creatinine clearance equation | 3 years
  Compare new estimated creatinine clearance equation for Taiwanese with Cockcroft-Gault equation

SECONDARY OUTCOMES:
Differences of daily urine creatinine excretion between Caucasian and Taiwanese | 3 years

OTHER OUTCOMES:
In which subgroup that difference between CG and MDRD is smallest or largest | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Fe-Lin Lin, Principal Investigator — National Taiwan University Hospital